CLINICAL TRIAL: NCT04211480
Title: an Open Label Trial of Evaluation of the Safety and Efficacy of Treatment With γ-globin Reactivated Autologous Hematopoietic Stem Cells in Subjects With β-thalassemia Major
Brief Title: Safety and Efficacy Evaluation of γ-globin Reactivated Autologous Hematopoietic Stem Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: Xiangya Hospital of Central South University (Other); The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-BRL-00CH1
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: β Thalassemia Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- γ-globin reactivated autologous hematopoietic stem cells (Experimental): each subject will accept one dose of γ-globin reactivated autologous hematopoietic stem cells
  Interventions: Biological: γ-globin reactivated autologous hematopoietic stem cells

INTERVENTIONS:
Biological: γ-globin reactivated autologous hematopoietic stem cells — gene edited autologous hematopoietic stem cells with γ-globin expression

SUMMARY:
This is a non-randomized, open label, single-dose, phase 1/2 study in up to 12 participants with β-thalassemia major.This study aims to evaluate the safety and efficacy of the treatment with γ-globin reactivated autologous hematopoietic stem cells in subjects with β-thalassemia major.

DETAILED DESCRIPTION:
γ-globin reactivated autologous hematopoietic stem cells will be manufactured using Crispr/Cas9 gene editing system. Subject participation for this study will be 1 year. Subjects who enroll in this study will be asked to participate in a subsequent long-term follow up study that will monitor the safety and efficacy of the treatment they receive for up to 15 years post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand and voluntarily sign informed consent. 5-15years old. At least one legal guardian and/or Subjects to sign informed consent.
* Clinically diagnosed as β-thalassemia major, phenotypes including β0β0, β+β0,βEβ0 genotype.
* Subjects with no affection with EBV, HIV, CMV, TP, HAV, HBV and HCV.
* Subjects body condition eligible for autologous stem cell transplant.

Exclusion Criteria:

* Subjects acceptable for allogeneic hematopoietic stem cell transplantation and have an available fully matched related donor.
* Active bacterial, viral, or fungal infection.
* Treated with erythropoietin prior 3 months.
* Immediate family member with any known hematological tumor.
* Subjects with severe psychiatric disorders to be unable to cooperate.
* Recently diagnosed as malaria.
* History of complex autoimmune disease.
* Persistent aspartate transaminase (AST), alanine transaminase (ALT), or total bilirubin value >3 X the upper limit of normal (ULN).
* Subjects with severe heart, lung and kidney diseases.
* With serious iron overload, serum ferritin>5000mg/ml.
* Any other condition that would render the subject ineligible for HSCT, as determined by the attending transplant physician or Investigator.
* Subjects who are receiving treatment from another clinical study, or have received another gene therapy.
* Subjects or guardians had resisted the guidance of the attending doctor.
* Subjects whom the investigators do not consider appropriate for participating in this clinical study.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Safety evaluation of γ-globin reactivated autologous hematopoietic stem cells | up to 24 months post transplant
  Proportion of subjects with engraftment; Overall survival.
Incidence and severity of adverse events as a measure of safety and tolerability. Adverse events assessed according to NCI-CTCAE v5.0 criteria | up to 24 months post transplant
  Incidence of AEs and SAEs post transplant

SECONDARY OUTCOMES:
Efficacy evaluation of γ-globin reactivated autologous hematopoietic stem cells | up to 24 months post transplant
  Proportion of subjects achieving transfusion independence for at least 6 months (TI6); Proportion of subjects achieving TI12; Proportion of alleles with intended genetic modification in bone marrow cells; Change in total hemoglobin concentration; Change from baseline in annualized frequency and volume of packed RBC transfusions.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Fu, Prof., Principal Investigator — Xiangya Hospital Central University
Locations (1):
- Shanghai Bioray Laboratories Inc., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in published article will be shared, after deidentification (text, tables,figures and appendices). Other available documents include study protocol.
Supporting Information: Study Protocol
Time Frame: IPD sharing will begin at 6 months and end at 36 months following article publication.
Access Criteria: IPD will be shared with investigators for individual data meta-analysis, after their proposed use of the data has been approved by an independent review committee. Proposals should be directed to yxwu@bio.ecnu.edu.cn and fu.bin@csu.edu.cn. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Fu B, Liao J, Chen S, Li W, Wang Q, Hu J, Yang F, Hsiao S, Jiang Y, Wang L, Chen F, Zhang Y, Wang X, Li D, Liu M, Wu Y. CRISPR-Cas9-mediated gene editing of the BCL11A enhancer for pediatric beta0/beta0 transfusion-dependent beta-thalassemia. Nat Med. 2022 Aug;28(8):1573-1580. doi: 10.1038/s41591-022-01906-z. Epub 2022 Aug 4. PMID 35922667
- [Derived] Brusson M, Miccio A. Genome editing approaches to beta-hemoglobinopathies. Prog Mol Biol Transl Sci. 2021;182:153-183. doi: 10.1016/bs.pmbts.2021.01.025. Epub 2021 Mar 1. PMID 34175041